CLINICAL TRIAL: NCT00513604
Title: A Phase II Study Using Short-Term Cultured Anti-Tumor Autologous Lymphocytes Following a Lymphocyte Depleting Regimen in Metastatic Melanoma
Brief Title: Phase II Study of Short-Term Cultured Anti-Tumor Autologous Lymphocytes After Lymphocyte-Depleting Chemotherapy in Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Dr. Steven Rosenberg, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070176; 07-C-0176
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Melanoma; Malignant Melanoma; Melanoma, Experimental; Experimental Melanomas
Keywords: Clinical Response; Immunotherapy; Cancer; Cytokines; Adoptive Cell Therapy; Melanoma; Skin Cancer; Malignant Melanoma
MeSH Terms: conditions — Melanoma; Melanoma, Experimental; Neoplasms; Skin Neoplasms | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 - NMA, TIL, aldesleukin (Experimental): Cohort 1 - Nonmyeloablative (NMA), tumor infiltrating lymphocytes (TIL), & high dose (HD) aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by bulk young tumor infiltrating lymphocytes and high dose aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. Bulk young TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
  Cohort 1 = unselected TIL
  Interventions: Biological: aldesleukin; Biological: therapeutic autologous lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine phosphate
- Cohort 2 - NMA, CD4+ TIL, aldesleukin (Experimental): Cohort 2 - Nonmyeloablative (NMA), cluster of differentiation 4 (CD4+) depleted tumor infiltrating lymphocytes (TIL), aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by CD4+ depleted tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
  Cohort 2 = CD4+ depleted (selected) TIL
  Interventions: Biological: aldesleukin; Biological: therapeutic autologous lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine phosphate
- Cohort 3 - NMA, total body irradiation (Experimental): Cohort 3 - Nonmyeloablative (NMA), total body irradiation (TBI):
  Nonmyeloablative chemotherapeutic conditioning regimen and 2 gray units (Gy) of total body irradiation followed by cluster of differentiation 4 (CD4+) depleted tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL 2Gy (gray units) of total body irradiation (TBI) twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute using a linear accelerator in Radiation Oncology Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
  Cohort 3 = CD4 + depleted (selected) TIL + 600Gy radiation
  Interventions: Biological: aldesleukin; Biological: therapeutic autologous lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine phosphate; Radiation: Total body irradiation
- Cohort 4 - NMA, young TIL, aldesleukin (Experimental): Cohort 4 - Nonmyeloablative (NMA), tumor infiltrating lymphocytes (TIL), aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by bulk young tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. Bulk young TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
  Cohort 4 = unselected TIL - it is the SAME as cohort 1
  Interventions: Biological: aldesleukin; Biological: therapeutic autologous lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine phosphate
- Cohort 5 - NMA, CD4+TIL, HD aldesleukin (Experimental): Cohort 5 - Nonmyeloablative (NMA), cluster of differentiation 4 (CD4+) tumor infiltrating lymphocytes (TIL), high dose (HD) aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by CD4+ depleted tumor infiltrating lymphocytes and high dose aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
  Cohort 5 = CD4 + depleted TIL - it is the SAME as cohort 2
  Interventions: Biological: aldesleukin; Biological: therapeutic autologous lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin — Given subcutaneously every 8 hours for up to 15 doses, day 0, 720,000 IU/kg
  Other Names: IL-2
Biological: therapeutic autologous lymphocytes — Given as infusion, up to 3 x 10^11 lymphocytes (minimum of 1 x 10^9), day 0
Drug: Cyclophosphamide — Given intravenously 60 mg/kg/day, day -7 to -6
Drug: Fludarabine phosphate — Given intravenously 25 mg/m^2/day over 15-30 minutes, day -5 to -1
  Other Names: Fludara
Radiation: Total body irradiation — 600 cGy
  Other Names: TBI
  Arms: Cohort 3 - NMA, total body irradiation

SUMMARY:
Background:

* Most therapeutic therapies for metastatic melanoma have focused on the ability of T-cell lymphocytes to kill cells of tumors.
* An adaptive cell transfer therapy has been pioneered, in which cells are grown for a short time in the laboratory. The way they are grown may have a better effect in a patient's body than do other cells that are cultured for a longer time.

Objectives:

* To determine whether tumor-infiltrating lymphocytes (TIL) can be put in cells removed from patients' tumors or blood and then reinfused, with the purpose of shrinking tumors.
* To evaluate safety and effectiveness of the treatment.

Eligibility:

* Patients 18 years of age or older with metastatic cancer melanoma (cancer that has spread beyond the original site).
* Patient's leukocyte antigen type is human leukocyte antigens (HLA-A) 0201.

Design:

-Patients undergo the following procedures:

* Leukapheresis (on two occasions). This is a method of collecting large numbers of white blood cells. The cells obtained in the first leukapheresis procedure are grown in the laboratory, and the TIL cells (called young TIL cells) are inserted into the cells using an inactivated (harmless) virus in a process called retroviral transduction. Cells collected in the second leukapheresis procedure are used to evaluate the effectiveness of the study treatment.
* Chemotherapy. Patients are given chemotherapy through a vein (intravenously, IV) over 1 hour for 2 days to suppress the immune system so that the patient's immune cells do not interfere with the treatment.
* Treatment with young TIL cells. Patients receive an IV infusion of the treated cells, followed by infusions the drug aldesleukin-2 (IL-2), which helps boost the effectiveness of the treated white cells.
* Patients are given support medications to prevent complications such as infections.
* Patients may undergo a tumor biopsy (removal of a small piece of tumor tissue).
* Patients are evaluated with laboratory tests and imaging tests, such as computed tomography (CT) scans, 4 to 6 weeks after treatment and then once a month for 3 to 4 months to determine the response to treatment.
* Patients have blood tests at 3, 6, and 12 months and then annually for 5 years.

DETAILED DESCRIPTION:
Background:

* Tumor Infiltrating Lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered to an autologous patient with high dose (HD) IL-2 following a non-myeloablative (NMA) but lymphodepleting chemotherapy preparative regimen.
* Clinical investigations and preclinical animal models have demonstrated that less time in culture, longer telomeres, and a less differentiated lymphocyte phenotype are associated with TIL that are capable of mediating objective clinical responses and persisting long term in the host.
* Previous methods for generating TIL require screening for anti-tumor specificity using gamma-interferon (IFN) production by the TIL. However, in vitro screening depends on autologous tumor reagents that are often unavailable; and gamma-IFN release in vitro may not be the best correlate to in vivo efficacy. Additionally, this method necessitates long in vitro culture times (44 days), and therefore reduces the clonal heterogeneity of TIL cultures, and results in TIL cultures with shorter telomere lengths and phenotypes that are skewed toward a more differentiated phenotype.
* In Surgery Branch pre-clinical experiments, we evaluated a method for rapidly generating young TIL from melanoma tumors with optimal phenotypic characteristics.

Objectives:

* In cohort 1, to determine the ability of autologous TIL cells infused after minimal in vitro culture in conjunction with high dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting preparative regimen to mediate tumor regression in patients with metastatic melanoma.
* In cohort 2, to determine the ability of autologous cluster of differentiation 4 (CD4+) cell depleted TIL cells infused after minimal in vitro culture in conjunction with high dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting preparative regimen to mediate tumor regression in patients with metastatic melanoma.
* In cohort 3, to determine the ability of autologous CD4+ cell depleted TIL cells infused after minimal in vitro culture in conjunction with high dose aldesleukin following chemoradiation lymphoid depleting regimen to mediate complete tumor regression in patients with metastatic melanoma.
* In a prospective randomized fashion, to compare the ability of autologous TIL cells (cohort 4) and autologous CD4plus cell depleted TIL cells (cohort regimen, to mediate tumor regression, progression free survival, and overall survival in patients with metastatic melanoma.
* Evaluate the toxicity of these treatment regimens.
* Determine the rate of repopulation of the young TIL cells in treated patients and establish in vitro correlates of TIL cultures that mediate objective response and in vivo persistence.

Eligibility:

Patients who 18 years of age or older must have:

* Metastatic melanoma;
* Normal values for basic laboratory values.

Patients may not have:

* Received prior cell transfer therapy that included non-myeloablative or ablative chemotherapy;
* Concurrent major medical illnesses;
* Any form of immunodeficiency;
* Severe hypersensitivity to any of the agents used in this study;
* Contraindications for high dose IL-2 administration.

Design:

* Patients will undergo resection to obtain tumor for generation of autologous TIL cultures.
* Cohort 1:

  * All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m^2/day IV) on days -5 through -1.
  * On day 0 patients will receive the infusion of autologous TIL and then begin high-dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
  * Clinical and Immunologic response will be evaluated about 4-6 weeks after TIL infusion.
  * Using a small optimal two-stage Phase II design, initially 21 patients will be enrolled, and if two or more of the first 21 patients has a clinical response (partial response (PR) or complete response (CR)), accrual will continue to 41 patients, targeting a 20% goal for objective response. Cohort 1 will be closed with amendment D.
* Cohort 2 will be initiated with amendment D whereby CD4+ cells will be eliminated from the cultures, using the Miltenyi Clinimacs apparatus, prior to performing the rapid expansion of the young TIL cells. Patients in cohort 2 will receive CD4+ cell depleted young unselected TIL. Patients will also receive high dose IL-2 after non-myeloablative but lymphodepleting chemotherapy preparative regimen as described above for cohort 1. Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion. Using a small optimal two-stage Phase II design, initially 18 patients will be enrolled, and if three or more of the first 18 patients have a clinical response (PR or CR), accrual will continue to 35 patients, targeting a 30% goal for objective response. With the initiation of Cohort 3 with amendment H, patients will only be accrued to Cohort 2 if they are not eligible to receive 600 cGy due to prior radiation, or to inability to mobilize cluster of differentiation 34 (CD34+) cells. Also at this time, accrual will be expanded to a total of 50 patients in cohort 2. Cohort 2 will be closed with amendment K.
* Cohort 3 will be initiated with amendment H, whereby patients will receive a chemoradiation lymphocyte depleting preparative regimen consisting of cyclophosphamide, fludarabine, and 600 cGy total body irradiation followed by intravenous infusion of autologous CD4+ cell depleted young TIL plus IV high dose IL-2. Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion. Using a small optimal two-stage Phase II design, initially 26 patients will be enrolled, and if one or more of the first 26 patients have a complete response (CR), accrual will continue to 51 patients, targeting a 10% goal for complete response. Cohort 3 will be closed with amendment K.

Prospective randomization between cohorts 4 and 5:

* Cohort 4:

  * All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m^2/day IV) on days -5 through -1.
  * On day 0 patients will receive the infusion of autologous TIL and then begin high-dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
  * Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion.
* Cohort 5

  * All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m^2/day IV) on days -5 through -1.
  * On day 0 patients will receive the infusion of autologous CD4+ depleted TIL and then begin high-dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).
  * Clinical and immunologic response will be evaluated about 4-6 weeks after TIL infusion.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma with at least one lesion that is resectable for tumor infiltrating lymphocytes (TIL) generation.
2. Patients with one to three brain metastases are eligible (lesions greater than or equal to 1 cm each, or symptomatic lesions must have been treated and stable for 3 months).
3. Greater than or equal to 18 years of age .
4. Willing to practice birth control during treatment and for four months after receiving the preparative regimen.
5. Life expectancy of greater than three months.
6. Willing to sign a durable power of attorney.
7. Able to understand and sign the Informed Consent Document.
8. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
9. Hematology:

   * Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim.
   * Normal white blood cell (WBC) (greater than 3000/ mm^3).
   * Hemoglobin greater than 8.0 g/dl.
   * Platelet count greater than 100,000/ mm^3.
10. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B or hepatitis C.
11. Chemistry: . Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal. Serum creatinine less than or equal to 1.6 mg/dl. Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.
12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
13. Six weeks must have elapsed since prior MDX-010 (Ipilimumab) therapy to allow antibody levels to decline.
14. Patients who have previously received any anti-CTLA4 (cytotoxic T-lymphocyte antigen 4) antibody and experienced treatment related colitis must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Prior cell transfer therapy that included non-myeloablative or ablative chemotherapy (for cohorts 4 and 5).
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Systemic steroid therapy required.
4. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
5. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and Acquired Immune Deficiency Syndrome (AIDS)).
6. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
10. Documented LVEF of less than or equal to 45% tested in patients with:

    - Clinically significant atrial and/or ventricular arrhythmias including but not limited to:

    atrial fibrillation, ventricular tachycardia, second or third degree heart block.

    - Age greater than or equal to 60 years old.
11. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking
    * Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2007-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Atkins MB, Kunkel L, Sznol M, Rosenberg SA. High-dose recombinant interleukin-2 therapy in patients with metastatic melanoma: long-term survival update. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S11-4. PMID 10685652
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- [Background] Rosenberg SA, Yannelli JR, Yang JC, Topalian SL, Schwartzentruber DJ, Weber JS, Parkinson DR, Seipp CA, Einhorn JH, White DE. Treatment of patients with metastatic melanoma with autologous tumor-infiltrating lymphocytes and interleukin 2. J Natl Cancer Inst. 1994 Aug 3;86(15):1159-66. doi: 10.1093/jnci/86.15.1159. PMID 8028037
- [Derived] Dudley ME, Gross CA, Somerville RP, Hong Y, Schaub NP, Rosati SF, White DE, Nathan D, Restifo NP, Steinberg SM, Wunderlich JR, Kammula US, Sherry RM, Yang JC, Phan GQ, Hughes MS, Laurencot CM, Rosenberg SA. Randomized selection design trial evaluating CD8+-enriched versus unselected tumor-infiltrating lymphocytes for adoptive cell therapy for patients with melanoma. J Clin Oncol. 2013 Jun 10;31(17):2152-9. doi: 10.1200/JCO.2012.46.6441. Epub 2013 May 6. PMID 23650429
- [Derived] Yao X, Ahmadzadeh M, Lu YC, Liewehr DJ, Dudley ME, Liu F, Schrump DS, Steinberg SM, Rosenberg SA, Robbins PF. Levels of peripheral CD4(+)FoxP3(+) regulatory T cells are negatively associated with clinical response to adoptive immunotherapy of human cancer. Blood. 2012 Jun 14;119(24):5688-96. doi: 10.1182/blood-2011-10-386482. Epub 2012 May 3. PMID 22555974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note with amendment K patients cohorts 1-3 were closed and patients were randomized between cohorts 4 and 5.
  The difference in the cohorts is NOT aldesleukin. The aldesleukin, cyclophosphamide and fludarabine are the same for each cohort. The difference is in the TIL and in cohort 3, the addition of radiation.
Groups:
- Cohort 1 - NMA, TIL, Aldesleukin: Cohort 1 - Nonmyeloablative (NMA), tumor infiltrating lymphocytes (TIL), & high dose (HD) aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by bulk young tumor infiltrating lymphocytes and high dose aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. Bulk young TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
- Cohort 2 - NMA, CD4+ TIL, Aldesleukin: Cohort 2 - Nonmyeloablative (NMA), cluster of differentiation 4 (CD4+) depleted tumor infiltrating lymphocytes (TIL), aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by CD4+ depleted tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
- Cohort 3 - NMA, Total Body Irradiation: Cohort 3 - Nonmyeloablative (NMA), total body irradiation (TBI):
  Nonmyeloablative chemotherapeutic conditioning regimen and 2 gray units (Gy) of total body irradiation followed by cluster of differentiation 4 (CD4+) depleted tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL 2Gy (gray units) of total body irradiation (TBI) twice on day -2 and once on day -1 (total dose 6 Gy) at a rate of 0.07 Gy/minute using a linear accelerator in Radiation Oncology Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
- Cohort 4 - NMA, Young TIL, Aldesleukin: Cohort 4 - Nonmyeloablative (NMA), tumor infiltrating lymphocytes (TIL), aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by bulk young tumor infiltrating lymphocytes and high dose (HD) aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. Bulk young TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days.
- Cohort 5 - NMA, CD4+TIL, HD Aldesleukin: Cohort 5 - Nonmyeloablative (NMA), cluster of differentiation 4 (CD4+) tumor infiltrating lymphocytes (TIL), high dose (HD) aldesleukin:
  Nonmyeloablative chemotherapeutic conditioning regimen followed by CD4+ depleted tumor infiltrating lymphocytes and high dose aldesleukin.
  Cyclophosphamide 60 mg/kg intravenous (IV) daily x 2 days. Fludarabine 25 mg/m^2 intravenous (IV) daily x 5 days. CD4+ depleted TIL Aldesleukin 720,000 IU/kg intravenous (IV) (based on body weight) over 15 minutes every eight hours for up to 5 days
Period: Overall Study
Arm/Group | Cohort 1 - NMA, TIL, Aldesleukin | Cohort 2 - NMA, CD4+ TIL, Aldesleukin | Cohort 3 - NMA, Total Body Irradiation | Cohort 4 - NMA, Young TIL, Aldesleukin | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin
Started | 26 (Cohort 1 = unselected TIL) | 39 (Cohort 2 = CD4+ depleted (selected) TIL) | 24 (Cohort 3 = CD4+ depleted (selected) TIL + 600Gy radiation) | 34 (Cohort 4 = unselected TIL - it is the SAME as cohort 1) | 35 (Cohort 5 = CD4+ depleted TIL-it is the SAME as cohort 2)
Completed | 24 | 36 | 21 | 34 | 35
Not Completed | 2 | 3 | 3 | 0 | 0
Not completed — Not treated | 2 | 0 | 1 | 0 | 0
Not completed — Death during treatment | 0 | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - NMA, TIL, Aldesleukin | Cohort 2 - NMA, CD4+ TIL, Aldesleukin | Cohort 3 - NMA, Total Body Irradiation | Cohort 4 - NMA, Young TIL, Aldesleukin | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin | Total
Number analyzed (Participants) | 26 | 39 | 24 | 34 | 35 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 26 | 39 | 24 | 34 | 34 | 157
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.7) | 46.3 (11.0) | 43.2 (11.9) | 45.1 (11.3) | 43.9 (12.0) | 45.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 11 | 11 | 18 | 72
  Male | 16 | 17 | 13 | 23 | 17 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 39 | 24 | 34 | 35 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 26 | 39 | 24 | 34 | 35 | 158
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 39 | 24 | 34 | 35 | 158

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical response is defined as complete response (CR)- a disappearance of all target lesions, partial response (PR) - at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression (PD)- at least a 20% increase in the sum of the LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: every 1-3 months until disease progression. Total length of time -8/7/2007 to 9/27/2012
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - NMA, TIL, Aldesleukin | Cohort 2 - NMA, CD4+ TIL, Aldesleukin | Cohort 3 - NMA, Total Body Irradiation | Cohort 4 - NMA, Young TIL, Aldesleukin | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin
Number analyzed (Participants) | 26 | 39 | 24 | 34 | 35
Participants
  Complete Response | 1 | 3 | 3 | 2 | 3
  Partial Response | 3 | 18 | 7 | 10 | 4
  Progression | 20 | 16 | 12 | 21 | 24
  Stable Disease | 0 | 0 | 0 | 1 | 4
  Not evaluable - cell product did not grow | 2 | 0 | 1 | 0 | 0
  Not evaluable-toxicities re:disease/death | 0 | 2 | 0 | 0 | 0
  Not evaluable - Patient died of sepsis | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 5 years
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - NMA, TIL, Aldesleukin | Cohort 2 - NMA, CD4+ TIL, Aldesleukin | Cohort 3 - NMA, Total Body Irradiation | Cohort 4 - NMA, Young TIL, Aldesleukin | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin
Number analyzed (Participants) | 26 | 39 | 24 | 34 | 35
Participants | 24 | 39 | 23 | 34 | 35

ADVERSE EVENTS:
Arm/Group | Cohort 1 - NMA, TIL, Aldesleukin | Cohort 2 - NMA, CD4+ TIL, Aldesleukin | Cohort 3 - NMA, Total Body Irradiation | Cohort 4 - NMA, Young TIL, Aldesleukin | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin
Serious Adverse Events (participants affected / at risk) | 9/26 | 8/39 | 5/24 | 5/34 | 4/35
Other Adverse Events (participants affected / at risk) | 24/26 | 39/39 | 23/24 | 34/34 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - NMA, TIL, Aldesleukin (N=26) | Cohort 2 - NMA, CD4+ TIL, Aldesleukin (N=39) | Cohort 3 - NMA, Total Body Irradiation (N=24) | Cohort 4 - NMA, Young TIL, Aldesleukin (N=34) | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders _ Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - NMA, TIL, Aldesleukin (N=26) | Cohort 2 - NMA, CD4+ TIL, Aldesleukin (N=39) | Cohort 3 - NMA, Total Body Irradiation (N=24) | Cohort 4 - NMA, Young TIL, Aldesleukin (N=34) | Cohort 5 - NMA, CD4+TIL, HD Aldesleukin (N=35)
Anemia (Blood and lymphatic system disorders) | 15 (17) | 27 (32) | 20 (23) | 11 (14) | 18 (21)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (10) | 17 (17) | 11 (11) | 14 (14) | 16 (16)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Chills (General disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 14 (17) | 9 (10) | 8 (8) | 10 (10)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter-related infection (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 10 (11) | 6 (7) | 7 (7) | 8 (8)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 5 (5) | 1 (1) | 3 (3) | 3 (3)
Creatinine increased (Investigations) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Electrocardiogram QT corrected interval prolong (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 24 (27) | 36 (40) | 23 (26) | 34 (37) | 35 (36)
Neutrophil count decreased (Investigations) | 24 (26) | 36 (41) | 23 (25) | 33 (34) | 35 (35)
Platelet count decreased (Investigations) | 21 (22) | 34 (37) | 23 (24) | 32 (32) | 31 (31)
Urine output decreased (Investigations) | 5 (5) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 14 (26) | 36 (37) | 22 (22) | 33 (33) | 35 (35)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (14) | 10 (11) | 5 (5) | 7 (8) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (7) | 4 (4) | 4 (5) | 4 (5) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (9) | 4 (5) | 0 (0) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 3 (3) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (9) | 7 (9) | 7 (8) | 10 (10) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 11 (12) | 4 (4) | 2 (3) | 4 (4)
peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 7 (7) | 9 (9) | 6 (6) | 7 (7) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 29 (29) | 11 (13) | 18 (18) | 9 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 17 (17) | 4 (4) | 9 (9) | 6 (6)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9) | 4 (4) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 10 (10) | 7 (7) | 2 (4) | 7 (7) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood and lymphatic system disorders _ Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (8) | 2 (2) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 13 (15) | 8 (9) | 7 (7) | 5 (5)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palmer-plantar erythrodyesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 16 (17) | 11 (11) | 6 (6) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No